CLINICAL TRIAL: NCT05995587
Title: Mindfulness-Based Cognitive Therapy in Managing Depressive Symptoms in Older People: A Non-Randomised Controlled Trial
Brief Title: Mindfulness-Based Cognitive Therapy in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Christian Family Service Centre (Other); The Mental Health Association of Hong Kong (Other); The Salvation Army, Hong Kong and Macau Command (Other); Caritas Medical Centre, Hong Kong (Other); Haven of Hope Hospital (Other)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA220105
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Depressive Symptoms
Keywords: Mindfulness-based cognitive therapy
MeSH Terms: conditions — Depression | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will either receive mindfulness training from a certified mindfulness teacher or from social workers (supervised by a certified mindfulness teacher). The care as usual group will receive usual service provided in District Elderly Community Centres (DECC) and Integrated Community Centre for Mental Wellness (ICCMW).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBCT (mindfulness teacher) (Experimental): Participants in the MBCT (mindfulness teacher) group will receive mindfulness training from a certified mindfulness teacher.
  Interventions: Behavioral: Mindfulness-based cognitive therapy (MBCT)
- MBCT (social workers) (Experimental): Participants in the MBCT (social workers) group will receive mindfulness training from social workers (supervised by a certified mindfulness teacher).
  Interventions: Behavioral: Mindfulness-based cognitive therapy (MBCT)
- Care as usual group (No Intervention): The care as usual group will receive usual service provided in District Elderly Community Centres (DECC) and Integrated Community Centre for Mental Wellness (ICCMW).

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy (MBCT) — MBCT combines mindfulness meditation with cognitive behavioural therapy (CBT) elements to reduce or prevent recurrent major depressive disorders.
  Arms: MBCT (mindfulness teacher); MBCT (social workers)

SUMMARY:
Mindfulness-based interventions, such as mindfulness-based cognitive therapy (MBCT), have the potential in improving psychological health in older people. With the growing older people population, there is a need for greater social welfare capacity to promote their well-being. The project aims to:

1. Evaluate the effectiveness of MBCT in improving mental health and mindfulness in older people with depressive symptoms as compared to care as usual;
2. Compare the effectiveness between MBCT led by mindfulness teacher and that led by social workers;
3. Examine psychological flexibility as a potential mechanism of change in MBCT for depressive symptoms.

DETAILED DESCRIPTION:
Depression is one of the most common yet under-recognized mental disorders in older adults in Hong Kong, and it is estimated that approximately one in 10 older people has clinically significant depression. With population aging, the number of older people with depression is slated to double in the next two decades, creating a substantial burden on the individuals, caregivers, and health care system. While pharmacological interventions are effective in reducing depression, medical risks can be complicated due to polypharmacy in older people. Non-pharmacological interventions may benefit the population by addressing the underlying dysfunctional cognitive processes associated with depression.

Mindfulness-based interventions, such as mindfulness-based cognitive therapy (MBCT), have the potential in improving psychological health in older people. MBCT is a group intervention originally designed to prevent recurrent depressive disorders. It combines mindfulness practices and cognitive-behavioural elements to enhance an individual's understanding of the interacting relationships among thoughts, emotions, bodily sensations, and behaviours. Mindfulness practice emphasizes on developing a moment-to-moment, non-judgmental awareness and may be helpful in alleviating depression by directing individual's attention to the present instead of ruminating in the past. Systematic reviews have shown the efficacy of MBCT in reducing depression, anxiety, loneliness, stress, sleep problems, ruminations, general mood, and positive affect. However, over half of the included studies lacked a control group and mixed findings were observed possibly because of inconsistent modifications to the protocol, methodological flaws, and study limitations.

The application of MBCT in the Chinese older population is understudied. Recently, a randomized controlled trial on MBCT for older people were conducted in Hong Kong. By comparing a standard MBCT to an active control group (physical exercise + health education) for older people with depression, it has been found that while both groups showed a reduction in the severity of depressive symptoms, only the MBCT group showed improvement in mindfulness.

With these promising findings, more studies are needed to establish the evidence base for the intervention and inform clinical practice in this population. The investigators aim to explore whether a modified MBCT based on older people's feedback can reduce depressive symptoms and improve mindfulness. With the growing older people population and thus a need for greater social welfare capacity to promote their well-being, the investigators will also examine whether a modified MBCT led by social workers under the supervision of a mindfulness teacher can benefit the population.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* have depressive symptoms of mild level or above, as indicated by scoring 5 or more in PHQ-9
* can give informed consent to participate

Exclusion Criteria:

* known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia
* imminent suicidal risk
* difficulty in communication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression at Week 8 | Baseline and Week 8
  Depression will be measured by the validated Chinese version of the Patient Health Questionnaire (PHQ-9). The total score will be used, ranging from 0 to 27. Higher scores indicate higher levels of depressive symptoms.
Change from baseline anxiety at Week 8 | Baseline and Week 8
  Anxiety will be measured by the validated Chinese version of the Generalized Anxiety Disorder scale (GAD-7). The total score will be used, ranging from 0 to 21. Higher scores indicate higher levels of anxiety symptoms.
Change from baseline stress at Week 8 | Baseline and Week 8
  Stress will be measured by the Chinese validated Perceived Stress Scale (PSS). The total score will be used, ranging from 0 to 40. Higher scores indicate greater stress.
Change from baseline mindfulness at Week 8 | Baseline and Week 8
  Mindfulness will be measured by the Chinese validated Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF). The total score of the FFMQ-SF (ranging from 20 to 100) as well as the total score (ranging from 4 to 20) of the five subscales (i.e., observe, describe, acting with awareness, nondjuding, and nonreactivity) will be used. Higher scores indicate higher mindfulness.
Change from baseline psychological flexibility at Week 8 | Baseline and Week 8
  Psychological flexibility will be assessed by the Chinese version of the Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT). Items are rated on a 0 (strongly disagree) to 6 (strongly agree) scale. The total score of the CompAct scale (ranging from 0 to 48), Valued Action subscale (ranging 0 to 18), Openness to Experience subscale (ranging from 0 to 18), and Behavioural Awareness subscale (ranging from 0 to 12) will be used. Higher scores indicate greater psychological flexibility.

OTHER OUTCOMES:
Change from baseline depression at Week 12 | Baseline and Week 12
  Depression will be measured by the validated Chinese version of the Patient Health Questionnaire (PHQ-9). The total score will be used, ranging from 0 to 27. Higher scores indicate higher levels of depressive symptoms.
Change from baseline anxiety at Week 12 | Baseline and Week 12
  Anxiety will be measured by the validated Chinese version of the Generalized Anxiety Disorder scale (GAD-7). The total score will be used, ranging from 0 to 21. Higher scores indicate higher levels of anxiety symptoms.
Change from baseline stress at Week 12 | Baseline and Week 12
  Stress will be measured by the Chinese validated Perceived Stress Scale (PSS). The total score will be used, ranging from 0 to 40. Higher scores indicate greater stress.
Change from baseline mindfulness at Week 12 | Baseline and Week 12
  Mindfulness will be measured by the Chinese validated Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF). The total score of the FFMQ-SF (ranging from 20 to 100) as well as the total score (ranging from 4 to 20) of the five subscales (i.e., observe, describe, acting with awareness, nondjuding, and nonreactivity) will be used. Higher scores indicate higher mindfulness.
Change from baseline psychological flexibility at Week 12 | Baseline and Week 12
  Psychological flexibility will be assessed by the Chinese version of the Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT). Items are rated on a 0 (strongly disagree) to 6 (strongly agree) scale. The total score of the CompAct scale (ranging from 0 to 48), Valued Action subscale (ranging 0 to 18), Openness to Experience subscale (ranging from 0 to 18), and Behavioural Awareness subscale (ranging from 0 to 12) will be used. Higher scores indicate greater psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Lum, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong; Gloria Wong, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong
Locations (6):
- Hong Kong (6):
  - Amity Place (Kwun Tong Central), Kwun Tong
  - Shun On District Elderly Community Centre (DECC), Kwun Tong
  - Haven of Hope District Elderly Community Service, Sai Kung
  - Wellness Zone - Integrated Community Centre for Mental Wellness, Sai Kung
  - Caritas Cheng Shing Fung District Elderly Centre (Sham Shui Po), Sham Shui Po
  - Tai Po Multi-service Centre for Senior Citizens, Tai Po

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geiger PJ, Boggero IA, Brake CA, Caldera CA, Combs HL, Peters JR, Baer RA. Mindfulness-Based Interventions for Older Adults: A Review of the Effects on Physical and Emotional Well-being. Mindfulness (N Y). 2016 Apr;7(2):296-307. doi: 10.1007/s12671-015-0444-1. Epub 2015 Sep 14. PMID 27200109
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Ng SM. Validation of the 10-item Chinese perceived stress scale in elderly service workers: one-factor versus two-factor structure. BMC Psychol. 2013 Jun 19;1(1):9. doi: 10.1186/2050-7283-1-9. eCollection 2013. PMID 25566361
- [Background] Shih VWY, Chan WC, Tai OK, Wong HL, Cheng CPW, Wong CSM. Mindfulness-Based Cognitive Therapy for Late-Life Depression: a Randomised Controlled Trial. East Asian Arch Psychiatry. 2021 Jun;31(2):27-35. doi: 10.12809/eaap2075. PMID 34987115
- [Background] Sun WJ, Xu L, Chan WM, Lam TH, Schooling CM. Depressive symptoms and suicide in 56,000 older Chinese: a Hong Kong cohort study. Soc Psychiatry Psychiatr Epidemiol. 2012 Apr;47(4):505-14. doi: 10.1007/s00127-011-0362-z. Epub 2011 Mar 8. PMID 21384121
- [Background] Tong X, An D, McGonigal A, Park SP, Zhou D. Validation of the Generalized Anxiety Disorder-7 (GAD-7) among Chinese people with epilepsy. Epilepsy Res. 2016 Feb;120:31-6. doi: 10.1016/j.eplepsyres.2015.11.019. Epub 2015 Nov 28. PMID 26709880
- [Background] Wang W, Bian Q, Zhao Y, Li X, Wang W, Du J, Zhang G, Zhou Q, Zhao M. Reliability and validity of the Chinese version of the Patient Health Questionnaire (PHQ-9) in the general population. Gen Hosp Psychiatry. 2014 Sep-Oct;36(5):539-44. doi: 10.1016/j.genhosppsych.2014.05.021. Epub 2014 Jun 6. PMID 25023953
- [Background] Thomas, R., Chur-Hansen, A. & Turner, M. A Systematic Review of Studies on the Use of Mindfulness-Based Cognitive Therapy for the Treatment of Anxiety and Depression in Older People. Mindfulness 11, 1599-1609 (2020). https://doi.org/10.1007/s12671-020-01336-3
- [Background] Morris, J. (2019). Development and validation of a short form of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT-SF). University of Nottingham.
- [Background] Segal, Z. V., Williams, J. M. G., & Teasdale, J. D. (2012). Mindfulness-based cognitive therapy for depression. Guilford Press.
- [Derived] Wang YH, Wang YL, Leung DKY, Ng ZLY, Chan OLH, Wong SMY, Chan RCL, Liu T, Wong GHY, Lum TYS. Effectiveness of an age-modified mindfulness-based cognitive therapy (MBCT) in improving mental health in older people with depressive symptoms: a non-randomised controlled trial. BMC Complement Med Ther. 2025 Feb 26;25(1):81. doi: 10.1186/s12906-025-04781-6. PMID 40011881

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05995587/Prot_SAP_000.pdf